CLINICAL TRIAL: NCT02934659
Title: Prospective, Multi-Center, Single Arm, Pilot Study to Evaluate Symptom Relief in Subjects With Medial Knee Osteoarthritis Treated With the AtlasTM Knee System for Load Reduction
Brief Title: Atlas Knee System Clinical System Clinical Study (USA)
Acronym: Atlas-USA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moximed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP0003 (formerly 102347)
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Investigational (Experimental): Intervention - Atlas Knee System device for medial knee osteoarthritis
  Interventions: Device: Atlas(TM) Knee System

INTERVENTIONS:
Device: Atlas(TM) Knee System — The Atlas System is an extra-capsular knee implant designed to unload the medial knee.
  Other Names: Atlas System

SUMMARY:
The primary objective of this pilot study is to collect data on the safety and effectiveness of the Atlas Knee System in subjects with medial knee osteoarthritis through 24 months postoperative follow-up.

DETAILED DESCRIPTION:
This study is designed as a prospective, multicenter, open-label, single arm, pilot study. Eligible subjects with symptomatic osteoarthritis of the medial compartment of the knee will be enrolled in the study and will receive the Atlas Knee Implant. The study population will consist of adult subjects age 25 to 80 years, with a diagnosis of medial knee osteoarthritis (Kellgen and Lawrence Grades 1-4, except those with bony erosions) and has pain in the study knee demonstrated as an overall WOMAC pain score of ≥ 40 (scale 0-100).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects age 25 to 80 years at time of screening
2. Clinical symptoms (such as pain primarily localized to the medial aspect of the knee and generally exacerbated by weight bearing) and radiographic evidence of osteoarthritis in the medial compartment of the knee

   * Weight-bearing Fixed Flexion view is recommended to verify radiographic evidence of osteoarthritis
   * KL Grade 1-4, except those with bony erosion
3. Has pain in the study knee as demonstrated by a minimum score of 40 (scale 0-100) on the WOMAC pain questions in KOOS
4. Has failed at least six (6) months of non-operative treatment with continued osteoarthritis (OA) pain. Prior treatment is defined as treatment with at least one of the following interventions (listed on the AAOS Clinical Practice Guidelines on the Treatment of Osteoarthritis of the Knee Non-arthroplasty):

   * Lifestyle modification
   * Weight loss, if BMI ≥35
   * Pain relievers
   * Physical Therapy
   * Orthotics (Splints, Braces)
   * Intra-Articular (IA) corticosteroid injections.
5. Knee flexion ≥90⁰
6. Body Mass Index (BMI) of <35 or weight <300 lbs.
7. Subjects who are able to give voluntary written informed consent to participate in this clinical investigation
8. Subjects, who, in the opinion of the Clinical Investigator, are able to understand this clinical investigation, cooperate with the investigational procedures, and are willing to return for all the required post-treatment follow up visits.

Exclusion Criteria:

1. Clinical symptoms or radiographic evidence of osteoarthritis in the lateral compartment of the study knee defined as Kellgren & Lawrence (K&L) grade of > 1
2. Clinical symptoms or radiographic evidence of osteoarthritis in the patella-femoral compartment of the study knee defined as K&L grade ≥ 3
3. Clinical symptoms or radiographic evidence of osteoarthritis at the contralateral knee that would preclude activity of daily living, stair climbing, stair descending, or requires the use of an assist device
4. Tibial-femoral alignment of more than 10⁰ of varus, or more than 6⁰ of valgus, as measured using anatomical axis on a standing Hip-Knee-Ankle or long standing AP view X-ray OR Hip-Knee-Ankle alignment of more than 16⁰ of varus, or more than 0⁰ of valgus, as measured using mechanical axis on a standing Hip-Knee-Ankle AP view x-ray
5. Previous joint modifying surgery in the study knee within 12 months prior to planned surgery date such as ligament reconstruction, meniscus repair, cartilage transplantation, and microfracture
6. Arthroscopic surgeries for joint lavage, meniscectomy, chondral debridement, and loose body removal are excluded if within 3 months prior to planned surgery date;
7. Active infection, sepsis, osteomyelitis or history of septic arthritis in any joint;
8. Previous lateral meniscectomy >30% of the study knee
9. Previous patellar surgery in the study knee
10. Previous osteotomy or failed knee joint replacement in the study knee
11. Hyperextension >5⁰
12. Flexion contracture > 10⁰
13. Pathologic ligamentous or meniscal instability (Lachman > 1) as assessed by the Investigator;
14. Suspected or documented allergy or hypersensitivity to cobalt, chromium, iron, or nickel metals;
15. Rheumatoid arthritis, other forms of inflammatory joint disease or autoimmune disorder;
16. Paget's disease or metabolic disorders which may impair bone formation;
17. Known or suspected diagnosis of Osteomalacia;
18. Known or suspected diagnosis of Osteonecrosis;
19. Rapid joint destruction, marked bone loss or bone resorption apparent on x-ray;
20. Osteoporosis or radiolucency of the femoral or tibial cortex on x-ray suggestive of moderate to severe osteoporosis, pathologic fractures, or bone mineral density T score of > 2.5 Standard Deviation (SD) below young adult reference mean (all subjects will be screened for risk of osteoporosis using the validated Osteoporosis Self-Assessment Tool (OST) score, subjects with high risk will undergo a DEXA scan to determine eligibility;
21. Charcot's joint disease or other severe neurosensory deficits;
22. Vascular insufficiency, muscular atrophy, neuromuscular disease;
23. Immunologically suppressed or immunocompromised;
24. History of systemic steroid treatment, medication use that affects bone metabolism (such as chemotherapy) within the previous 6 months, or radiotherapy within the previous 6 months
25. Any significant medical condition including:

    * Diabetes mellitus requiring daily insulin therapy
    * Neuropathic pain or fibromyalgia, or any knee or other pain requiring chronic pain management
    * Advanced liver and kidney diseases
    * Congestive heart failure
    * Uncontrolled transient ischemic attack
    * Cancer
    * HIV (immunocompromised subject)
    * Radicular symptoms associated with lumbar spine pathology
    * Neurological disorders that result in gait disturbance
    * Restless leg syndrome
    * History of complex regional pain syndrome (Reflex Sympathetic Dystrophy (RSD); l. Significant psychiatric disorders (such as major depression, anxiety disorders, bipolar disorder, and schizophrenia); m. History or active substance and alcohol dependence and abuse (meeting standard diagnostic criteria described in the Diagnostic and Statistical Manual of Mental Disorders DSM-IV)
26. Other factors that the investigator feels would interfere with the participation and completion of the study:

    * Planned relocation
    * Litigation for or workers compensation for musculoskeletal injuries or disorders
    * Uncooperative subject
    * Or any other reason.
27. Pregnancy or planning to become pregnant
28. Subjects who are currently involved in any investigational drug or device trial or have been enrolled in such trials within the last 3 months
29. Prisoners or wards of the state.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this pilot study is the rate of individual subject success at 24 months. A subject will be declared a clinical success if all of the following conditions are met at the 24-month follow-up: | Change at 24 months relative to baseline
  1. Clinically significant improvement of at least 20% from baseline on the WOMAC pain questions in the KOOS questionnaire with a change of ≥10 points;
  2. Clinically significant improvement of at least 20% from baseline on the WOMAC function questions in the KOOS questionnaire with a change of ≥10 points;
  3. Maintenance of normal range of motion (ROM) defined as:
     (a) Knee flexion ≥ 90 degrees; and (b) Knee extension within 10 degrees of the "neutral" or zero degree position;
  4. No subsequent surgical intervention of the medial knee (including device failures requiring removal or revision); and no serious device-related adverse events;
  5. Maintenance of implant integrity as evaluated by radiographic assessment. a. Implant integrity will be assessed following the Atlas Image Evaluation Protocol (102345).

CONTACTS AND LOCATIONS:
Overall Officials: Rose Weinstein, Study Director — Moximed
Locations (9):
- United States (9):
  - Banner-University Medical Center Phoenix, Phoenix, Arizona
  - Orthropaedic Research Foundation, Greenwood, Indiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Hospital for Special Surgery (HSS), New York, New York
  - Duke University, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Houston Methodist, Houston, Texas
  - University of Virginia, Dept. of Orthopaedic Surgery, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No